CLINICAL TRIAL: NCT04989712
Title: The Impact of Different Exercise Timings on Blood Glucose Control and Cognition in Children and Adolescents Using the Freestyle Libre Continuous Glucose Monitoring System
Brief Title: MOReS Freestyle Libre Validation Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Shelly Coe, Senior Lecturer, Oxford Brookes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LGHC072021
Record Dates: First submitted 2021-07-13; First posted 2021-08-04 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Blood Glucose; Executive Function; Cognitive Change
Keywords: MVPA; Glucose; Cognition; Children; Adolescents

STUDY DESIGN:
Intervention Model Description: Randomised cross over design. Participants act as own controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 20 minutes MVPA (Experimental): 20 minutes of moderate to vigorous exercise at 50-80% maximum heart rate to be performed on a cycle ergometer 40 minutes from the start of the testing session following consumption of a glucose solution at 0 mins. Glucose readings from the FreeStyle Libre to be taken at 0 mins, 30 mins, 60 mins, 90 mins and 120 mins. Cognitive tests to be carried out before the glucose solution is administered at 0 mins and at the 120 min point.
  Interventions: Other: Exposure
- 4 x 5 mins MVPA (Experimental): 4 bouts of 5 minutes of moderate to vigorous exercise at 50-80% maximum heart rate to be performed on a cycle ergometer 30 minutes from the start of the testing session and repeated at 60 mins, 90 mins and 120 mins following consumption of a glucose solution at 0 mins. Glucose readings from the FreeStyle Libre to be taken at 0 mins, 30 mins, 60 mins, 90 mins and 120 mins. Cognitive tests to be carried out before the glucose solution is administered at 0 mins and at the 120 min point.
  Interventions: Other: Exposure
- Uninterrupted sitting - No exercise, sitting session (control). (Experimental): A sitting only exposure, glucose solution to be consumed at 0 mins.Glucose readings from the FreeStyle Libre to be taken at 0 mins, 30 mins, 60 mins, 90 mins and 120 mins. Cognitive tests to be carried out before the glucose solution is administered at 0 mins and at the 120 min point
  Interventions: Other: Exposure

INTERVENTIONS:
Other: Exposure — Participants randomised to one of the three exposures

SUMMARY:
To measure the effects of interrupting prolonged sitting with brief standing physical activity interventions on physical and cognitive performance, health and wellbeing in young people.

DETAILED DESCRIPTION:
Cross over randomised exposure response experimental study in 10 healthy children and adolescents, to measure the effects of interrupting prolonged sitting with brief standing physical activity interventions on their physical and cognitive performance, mobility, health and wellbeing. The study will assess the extent of the immediate and short-term effects of interrupting sitting with brief moderate-vigorous physical activity (MVPA) breaks compared to a sitting only condition.

Dietary analysis and metabolic and cognitive tests after acute exercise will be performed on the participants to compare the FreeStyle Libre responses between those with and without disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Young people aged 9-18 years old
* No significant current or previous medical history
* Are able to participate safely in the study's assessments and brief interrupted sitting moderate to vigorous physical activity (MVPA)

Exclusion Criteria:

* Those with uncontrolled epilepsy/seizures (stable epilepsy/on medication > 12 weeks)
* Those who have Type 1 and Type 2 diabetes or other glucose intolerance or on medication for such conditions
* Those who experience contraindications to physical training
* Those who are on any form of steroids, anti-anxiety/depression drugs, birth control, beta-blockers, statin, adrenaline, HIV or Hepatitis C medications (these medications can affect the readings during the oral glucose tolerance test)
* Those with known allergies to plasters

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Executive Functioning - Eriksen Flanker Task | Maximum of two weeks
  The main outcome will be change in executive functioning from the start to the end of the session using the Eriksen Flanker Task. The test measures selective attention and executive control and measures speed (milliseconds) and accuracy (number of responses correct). This will be performed before the oral glucose tolerance test and again at the end of each session.
Working Memory - WISC Digit Span | Maximum of two weeks
  Wechsler Intelligence Scale for Children (WISC) Digit Span will test attention and working memory. The total score is calculated by the number of correct responses. This will be performed before the oral glucose tolerance test and again at the end of each session.

SECONDARY OUTCOMES:
Oral Glucose Tolerance Test (OGTT) | Maximum of two weeks
  On arrival an OGTT, simulating insulin and glucose response comparable to that following a meal will be given. Children will follow an identical protocol for OGTT during all conditions. Children will be asked to fast the night before, for 10 hours prior to the test. They will arrive fasted, have a baseline glucose reading taken and will be given the OGTT, followed by sit only or sit in addition to physical activity breaks regimens. For the OGTT the stimulus is 1.75g/kg body weight of glucose solution. A Freestyle Libre glucose monitoring system will be placed on the participants' arm and glucose readings will be monitored at timed intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Dawes, PhD, Principal Investigator — Oxford Brookes University
Locations (1):
- Oxford Brookes University, Oxford, Oxfordshire, United Kingdom